CLINICAL TRIAL: NCT03532958
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Trial of Intravenous BNZ-1 in Patients With Moderate to Severe Alopecia Areata
Brief Title: Phase 2 Trial of BNZ-1 in Patients With Moderate to Severe Alopecia Areata
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Transfer of study sponsor
Sponsor: Equillium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNZ1-CT-204
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Normal saline
- Low Dose BNZ-1 (Experimental): 0.5 mg/kg QW
  Interventions: Drug: BNZ-1
- Moderate Dose BNZ-1 (Experimental): 2 mg/kg QW
  Interventions: Drug: BNZ-1

INTERVENTIONS:
Drug: BNZ-1 — PEGylated peptide inhibitor of IL-2, IL-9, and IL-15
  Arms: Low Dose BNZ-1; Moderate Dose BNZ-1
Drug: Normal saline — Dose volume consistent with weight-based dosing of BNZ-1
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multi-center, dose-ranging study to characterize the efficacy and safety of BNZ-1 administered by slow IV push weekly for 3 months to adults diagnosed with moderate to severe alopecia areata, defined as having a >50% loss of terminal hair on the scalp. The study has three periods:

* 30-Day Screening Period
* 3-Month Treatment Period
* 3-Month Follow-up Period The study will be conducted at approximately 15-20 clinical sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a diagnosis of moderate to severe AA defined as the presence of ≥50% total terminal hair loss at baseline as measured using the SALT score for > 6 months, but <10 yrs. Includes Alopecia Totalis and Alopecia Universalis
2. Patients may be naïve to treatment or have been treated with intralesional (IL) steroids or other treatments for AA, with a washout of at least 30 days or 5 times the elimination half-life prior to Day 1.
3. Prior treatment with a janus kinase (JAK) inhibitor (e.g., tofacitinib, ruxolitnib) is allowed, but patients considered refractory to a JAK inhibitor are excluded from this trial.

Exclusion Criteria:

e subjects from this study if any of the following criteria are met:

1. Clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, renal, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult, or that would put the subject at risk by participating in the study in the opinion of the Investigator. Other active dermatologic conditions, including but not limited to vitiligo, atopic dermatitis, or non-scalp psoriasis are not exclusionary.
2. Patients with active inflammatory skin disease on the scalp, including but not limited to psoriasis, seborrheic dermatitis or folliculitis, which cannot be adequately controlled prior to screening.
3. Ongoing treatment with an immune system modulator or suppressant that cannot be discontinued prior to screening and at least 30 days or 5-times the elimination half-life prior to treatment.
4. Any ongoing topical treatment for alopecia areata
5. History of or currently active primary or secondary immunodeficiency.
6. Known active bacterial, viral, fungal, mycobacterial infection, or other infection (including latent tuberculosis [TB] unless treatment is documented or atypical mycobacterial disease [but excluding fungal infection of nail beds, minor upper respiratory tract infection, and minor skin conditions]), or any major episode of infection that required hospitalization or treatment with IV antibiotics within 60 days of study drug administration or oral antibiotics within 30 days prior to study drug administration.
7. Received other investigational products or therapy in the 60 days prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline using the Severity of Alopecia Tool (SALT) score | 3 months
Treatment-Emergent Adverse Events | 3 months
  Safety profile defined as incidence, severity and relationship of treatment-emergent adverse events

SECONDARY OUTCOMES:
Alopecia Areata Investigator Global Assessment (AA-IGA) | 3 & 6 months
  Hair Satisfaction Scale
Patient Global Assessment | 3 & 6 months
  Hair satisfaction scale
Proportion of Patients with SALT50 | 3 months & 6 months
Proportion of Patients with SALT75 | 3 months & 6 months
Proportion of Patients with SALT90 | 3 months & 6 months
Proportion of Patients with SALT100 (Disease-free) | 3 months & 6 months
Change from Baseline on Alopecia Areata Symptom Impact Scale (AASIS) | 3 months
Change from Baseline on Dermatology Life Quality Index (DLQI) | 3 months

IPD SHARING:
Plan to Share IPD: Undecided